CLINICAL TRIAL: NCT06596356
Title: A Phase 1 Mass Balance Study of TS-172 in Healthy Adult Subjects
Brief Title: A Mass Balance Study of TS-172 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS172-02-02
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-11

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C] TS-172 (Experimental): Participants will receive oral [14C] TS-172 under fasted conditions
  Interventions: Drug: [14C] TS-172

INTERVENTIONS:
Drug: [14C] TS-172 — Subjects will receive single dose of about 30 mg of TS-172 containing 1 MBq [14C]TS-172 as an oral solution

SUMMARY:
To assess the plasma pharmacokinetics, the routes extent of elimination, and the metabolites of TS-172 after single oral dose of [14C] TS-172 in Japanese healthy male subjects.

To assess the safety of single oral dose of [14C] TS-172 in Japanese healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males aged >=20 and <40 years at the signing of informed consent
* Subjects whose body mass index (BMI) >=18.5 and <25.0 kg/m2 at screening
* Subjects who have no abnormal findings in the physical examination, vital signs, and standard 12-lead ECG in the screening test and the test on the day of admission and the test obtained prior to administration of the investigational drug, and whose clinical test results are within the standard values of the clinical trial site in the screening test and the test on the day of admission. However, if who showed abnormal findings or values outside the reference ranges but not clinically significant, they can be enrolled in clinical trials based on comprehensive consideration of medical viewpoints by the principal investigator(s) or subinvestigator(s).
* Subjects who understand, and have willingness and ability to read and sign, the informed consent form

Exclusion Criteria:

* Subjects who have been administered substances labelled with radioisotopes or exposed to high levels of radiation (e.g. CT scan, gastric X-ray, PET scan) within one year prior to dosing of the investigational drug.
* Occupationally exposed worker within one year prior to dosing of the investigational drug (e.g. workers who handle nuclear power or radioactive substances)
* Subjects who have had 3 days or less that one or more spontaneous defecations (defecation that occurs without laxatives, enemas, disimpaction) within 7 days before consent is obtained or during the 7 days until on the day of admission. Those who have diarrhea during the 7 days until on the day of admission
* History of any disease or surgery which have impact on investigational drug absorption such as gastrointestinal ulcer, gastrectomy, gastroenterostomy or bowel resection

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration in whole blood and plasma | Up to 240 hours after dosing
Calculation of cumulative urinary and fecal recovery of total radioactivity, and calculation of mass balance as a sum of the percentages of total radioactivity recovered in urine and faeces | Up to 240 hours after dosing
Concentration of unchanged form and its major metabolites in plasma | Up to 240 hours after dosing
Percentage of unchanged form and metabolites to total radioactivity in plasma | Up to 240 hours after dosing
Percentage of unchanged form and metabolites to total radioactivity in urine and faeces | Up to 240 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No